CLINICAL TRIAL: NCT02486276
Title: The Effect of Sumatriptan and Placebo on Cilostazol Induced Headache. Development of a Pragmatic Migraine Model
Brief Title: The Effect of Sumatriptan and Placebo on Cilostazol Induced Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Emma Katrine Hansen, Medical doctor, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-8-2014-009
Record Dates: First submitted 2015-06-04; First posted 2015-07-01 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Cilostazol; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sumatriptan (Active Comparator): headache is induced with Cilostazol. This headache is treated double-blinded with 1 tablet of sumatriptan 50 mg
  Interventions: Drug: Cilostazol; Drug: Sumatriptan
- Placebo (Placebo Comparator): headache is induced with Cilostazol. This headache is treated double-blinded with 1 tablet of placebo
  Interventions: Drug: Cilostazol; Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol — Cilostazol is given both study days to induce headache. One day the headache is treated with placebo and the other day with sumatriptan
  Other Names: Pletal
Drug: Sumatriptan — Cilostazol is given both study days to induce headache. One day the headache is treated with placebo and the other day with sumatriptan
  Other Names: Imigran
  Arms: Sumatriptan
Drug: Placebo — Cilostazol is given both study days to induce headache. One day the headache is treated with placebo and the other day with sumatriptan
  Arms: Placebo

SUMMARY:
To develop a pragmatic migraine model the investigators will induce headache in healthy volunteers and in patients with migraine without aura with a phosphodiesterase inhibitor (cilostazol). If the headache responds to sumatriptan, the model can be used to test new drug candidates.

DETAILED DESCRIPTION:
There remains a great need for more effective anti-migraine drugs with fewer side effects. Human experimental models are valuable in early phase development of new anti-migraine drugs but useful models have not yet been developed. The investigators' group has shown that Cilostazol, a phosphodiesterase inhibitor induce headache/migraine in both healthy volunteers and in patients with migraine without aura (MO). To validate this model, the headache must respond to specific migraine treatment with sumatriptan.

Hypothesis: Cilostazol induces a migraine-like headache in both healthy subjects and in MO-patients and induced headache responds to a specific anti migraine drug; sumatriptan.

Aim: Developing a pragmatic and valid model for the testing of new anti-migraine drugs.

ELIGIBILITY:
Inclusion criteria:

Healthy:

* Healthy subjects of both sexes
* Age 18-70 years
* Weight 50-90 kg.
* Females were requested to use effective contraception.

Migraine patients:

* Migraine patients who meet IHS criteria for migraine with or without aura of both sexes
* 18-70 years
* 45-95 kg.

Exclusion Criteria:

Healthy:

* Any type of headache (except episodic tension-type headache < 1 day per week)
* Serious somatic or psychiatric disease
* Pregnancy
* Intake of daily medication (except oral contraceptives).

Migraine patients:

* Any other type of headache then migraine without aura (except episodic tension-type headache < 1 day per week)
* Serious somatic or psychiatric disease
* Pregnancy
* Intake of daily medication (except oral contraceptives)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Difference in median headache score 2 hours after sumatriptan/placebo | 2 hours
  The investigators will assess the outcome measures 1 year after the beginning of the study

SECONDARY OUTCOMES:
Area under the headache score curve | 12 hours
  The investigators will assess the outcome measures 1 year after the beginning of the study

CONTACTS AND LOCATIONS:
Overall Officials: Emma Katrine Hansen, Doctor, Principal Investigator — Danish Headache Center
Locations (1):
- Emma Katrine Hansen, Copenhagen, Glostrup, Denmark

REFERENCES:
- [Derived] Falkenberg K, Dunga BOA, Guo S, Ashina M, Olesen J. Cilostazol induced migraine does not respond to sumatriptan in a double blind trial. J Headache Pain. 2018 Feb 2;19(1):11. doi: 10.1186/s10194-018-0841-7. PMID 29396788